CLINICAL TRIAL: NCT03921697
Title: Parkinson App SmarTphone Aimed to Improve Walking Ability and Reduce Fall (P.A.S.T.A.)
Brief Title: Improving Walking Ability in Parkinson Disease
Acronym: PASTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Augusto Fusco, Principal Investigator; M.D.; Ph.D., Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: GR-2016-02362879
Record Dates: First submitted 2019-03-18; First posted 2019-04-19 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease
Keywords: Technological Rehabilitation; Digital Inclusion
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson Disease Patients: Patients with PD will be recruited at Fondazione Policlinico Universitario Gemelli and Fondazione Don Gnocchi ONLUS in Rome. All included patients will be affected by idiopathic PD. Clinical data will be acquired by a trained neurologist.
  We will remotely monitor 300 patients through wearable sensors. Subjects will be instructed to wear the sensor for 14 consecutive days.
  Interventions: Device: Werable sensors

INTERVENTIONS:
Device: Werable sensors — Parkinson Disease Patients monitored by werable sensors

SUMMARY:
Gait impairments of patients with Parkinson's disease (PD) limit the independence in the daily activities and sensibly increase the risk of falls. New gait analysis methods, based on wearable inertial sensors, have been proposed to track the gait features during treatment and in real-life conditions. Gait training based on auditory cues as Rhythmical Auditory Stimulation (RAS) have preliminarily shown positive effects improving gait velocity, stride length, step cadence of walking in PD. In the current project, the research group will aim to develop a smartphone application (Parkinson App Smartphone Aimed: P.A.St.A.) integrated with sensors and RAS. In a second time, investigators will analyze the spatio-temporal gait parameters obtained by the wearable sensors and the sociodemographic and clinical data, thus generating a big data set, to improve the knowledge about current pharmacological therapies and rehabilitation.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a chronic and progressive movement disorder, mainly due to an altered motor control. Gait impairments are the primary symptoms in patients with PD, with a decreased step length and walking speed, abnormal gait phases distribution, inconstant pace, gait asymmetry and reduced joint coordination. The postural instability and the deterioration of the gait features sensibly increase the risk of falls in these patients, resulting in loss of independence and a worsening of long-term prognosis. It has been clearly demonstrated that motor impairments are connected to a dysfunction of basal ganglia, a brain structure that works as a "pacemaker" for the activation (and deactivation) of each sub-movement within a repetitive movement sequence. Disruption of internal rhythmic cues in PD may explain the poor smoothness of the movement execution and the difficulties in regulating stride length, resulting in a cadence increase. Levodopa therapy is the most effective treatment to improve the symptoms in PD, but a long-term administration reduces its efficiency over time and it is responsible for collateral effects (dyskinesia). Hence, researches have investigated alternative non-pharmacological approaches, based on auditory cues as the Rhythmical Auditory Stimulation (RAS). A large number of studies have reported positive effects both after a single session of treatment and after longer training programs, with improved gait velocity, cadence, and stride length as well as in the symmetry of muscle activation for upper and lower extremities. In such studies, RAS frequencies are pre-set as percentages of the patient's preferred walking frequency. Because the duration of all the therapies may change over time, it is necessary a continuous adjustment of the dosage and type of treatment, based both on patients' monitoring of the symptoms and on objective evaluations. Gait analysis (GA) methods have been proposed and validated for the study of physiologic gait and in several diseases. The traditional systems of GA are based on optoelectronic systems, but they are expensive, not portable and requiring skilled operators. The assessment is always performed in laboratories with experimental set-ups, likely different from real-life walking (noise environments, presence of objects and people or unlevelled pavement, different colors).

Consequently, traditional GA is not reliable for the daily control of the treatments or for the assessment of the real-life situations. Recently, researchers have developed wearable systems, based on Inertial Measurement Units (IMUs). Even if a considerable number of studies have explored the validity of IMUs analysis, very few have been involved in PD motion analyses. During the last few years, a set of wearable devices embedding inertial sensors, are spread on the market as low-cost solutions for monitoring human motion activities. While, they still have to be fully validated in accuracy, these systems can provide the user information to track his/her own activity. This persuasive technology has a terrific potential to enhance physical activity and motivation of the patients, with the advantage of prolonged and continuous recording.

The use and the analyses of a large amount of objective data (big data set) is the new frontier for an efficient use of scientific time and resources, engaging the care coordination program, saving economic resources, and providing a higher quality of care. In addition, these systems, integrated with a web-based application, telemedicine and mobile smartphones, could help clinicians to address more properly the treatments through a real-time monitoring in an everyday life. Our research group has been involved in the clinical evaluation of different aspects of gait quality in many neurological conditions, PD included. Investigators have already shown as wearable accelerometers could be useful in the quantitative assessment of the dynamic gait stability, in correlation with clinical scores. Researchers have also found that accelerations could be altered in a pathology-specific manner (intellectual disabilities performing different tasks simultaneously). A similar condition can be observed also in PD, showing that only the intrinsic gait harmony significantly correlate with severity of gait impairments. In the recent years, a lot of wearable tools have become available to quantify the daily activity. This is particularly important for possible therapeutic use of the RAS, that is addressed to restore a harmonic pace in patients with PD.

Specific Aim 1: To analyze motor pattern in PD patients in real life setting, gait features will be obtained by wearable sensors in order to relate them with clinical and demographical data.

Specific Aim 2: To improve walking abilities and to reduce the risk of falls in patients with PD, researchers will test a real-time acoustic feed-back (RAS) and alerts from integrated sensors connected with a suitable and easy-to-use application for smartphones.

Specific Aim 3: To improve pharmacological and rehabilitative protocols, investigators will analyze the daily life gait and motility data and the clinical features to test the theoretical risk model of falls.

Experimental Design Aim 1: Patients with PD will be recruited at Fondazione Policlinico Universitario Gemelli and Fondazione Don Gnocchi ONLUS in Rome. All included patients will be affected by idiopathic PD. Clinical data will be acquired by a trained neurologist.

Three hundred patients will be remotely monitored through wearable sensors. Subjects will be instructed to wear the sensor for 14 consecutive days. Each patient will have more than 100 measurements every second, generating a large amount of data, which will be stored in a database and subsequently filtered for data of interest. Spatio-temporal gait parameterswill provide information to monitor the performance of patient's walking in order to get an accurate measure of the overall efficacy of the locomotor function. Then, they will be integrated with the electronic patient records. Clinical data, as physician's prescriptions, medical imaging and other administrative data will be recorded. Finally, a risk model for the prediction of falls will be constructed.

Experimental Design Aim 2: After the analysis of the obtained data, an application will be developed (Parkinson App Smartphone Aimed: P.A.St.A.), it will be characterized by reliability, easy-to-use, visual clarity, and affordability.

This application will be able to: 1) record the gait features sending them to a server in the cloud; 2) provide acoustic feedback adapted on patient's gait features (with higher or lower frequency on the basis of the patient's needs and on the predictive risks); 3) provide alert on the basis of risk indices (risk indices will be identified according to a risk model for the prediction of falls) and 4) be updated whenever needed (e.g. after a fall). Fifty patients will be provided with a smartphone, after a training on the use of the software application developed by the team project. They will use the application for a period of 14 consecutive days. Clinical assessments with scales will be performed, pre- and post-use of P.A.St.A., to analyze the motor function and the postural stability and, finally, the quality of life. In addition, the compliance to the adoption of the novel technology will be investigated.

Experimental Design Aim 3: The obtained computational data will be related with clinical features and gait patterns to identify clinical biomarkers for gait impairment in PD. The availability of a big data-sets, powered by the assessments of thousands of patients with PD, will allow the improvement of knowledge on motor pattern in real life setting and to improve the current therapeutic approach.

Metodologies and statistical analyses: All statistical analyses will be conducted using Stata software.

AIM 1 - Data will be summarized as frequencies and percentages for categorical variables. Continuous variables will be analyzed as means and standard deviations or medians and ranges. Investigators will look for normality by using normal plots or by significance tests (e.g. Shapiro-Wilk W test). The incidence of falls will be measured and the circumstances under which they occur and their consequences will be described, categorized as no injury, minor or major injuries. A multiple logistic regression analysis will be used to determine independent predictors of falls. Variables will be selected for entry into the logistic model based on the results of a univariate analyses. The Hosmer-Lemeshow goodnessof-fit test will be used to assess how well the model accounted for specific outcomes. The prediction model for falls will be developed from the results of the multivariate analysis. The predictive score will be calculated by odds ratio based scoring method, and the nearest integer scores will be assigned to each predictor. Model discriminative power will be evaluated by receiver-operating characteristic area under the curve analysis.

AIM 2 - Data recorded will be processed to extract gait and dynamic balance parameters. The incidence of falls, the use of RAS and its correlation to the risks indices within the 14 days of follow-up will be measured. The Wilcoxon signed-rank test will be performed to compare the number of fall(s) before and after the use of P.A.St.A.

AIM 3 - Spatio-temporal gait parameters, and demographic and clinical characteristics of patients before therapies, will be compared using the Chi squared test, Fisher's exact test, and independent t-tests where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease diagnosed by a neurologist
* Ability to sign informed consent

Exclusion Criteria:

* Inability to sign informed consent
* Inability to fill out questionnaires (i.e. due to poor vision, inability to read, etc)
* Presence of psychiatric diseases (episode or any form of psychosis, diagnosed by a psychiatrist in the last year).
* Age under 18 yrs old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients will be enrolled among outpatients of the Movement Disorders Unit of the Gemelli University Hospital and outpatients of the Fondazione Don Carlo Gnocchi Onlus.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlations between inertial sensor-derived measures of motor function and clinician ratings during performance of the UPDRS part 3 and total exam at baseline | Fourteen days
  Features extracted from continuous accelerometer signals recorded during real life for fourteen days, will be correlated with each relevant component of the UPDRS part 3 and corresponding clinician ratings to quantify the relationship between these measures.

SECONDARY OUTCOMES:
Time Up&Go | Baseline
  Time Up&Go is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require.

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Fusco, M.D.; Ph.D., Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- Fondazione Don Carlo Gnocchi Onlus, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubinstein TC, Giladi N, Hausdorff JM. The power of cueing to circumvent dopamine deficits: a review of physical therapy treatment of gait disturbances in Parkinson's disease. Mov Disord. 2002 Nov;17(6):1148-60. doi: 10.1002/mds.10259. PMID 12465051
- [Background] Rogers MW. Disorders of posture, balance, and gait in Parkinson's disease. Clin Geriatr Med. 1996 Nov;12(4):825-45. PMID 8890118
- [Background] Yogev G, Plotnik M, Peretz C, Giladi N, Hausdorff JM. Gait asymmetry in patients with Parkinson's disease and elderly fallers: when does the bilateral coordination of gait require attention? Exp Brain Res. 2007 Mar;177(3):336-46. doi: 10.1007/s00221-006-0676-3. PMID 16972073
- [Background] Heiderscheit BC. Movement Variability as a Clinical Measure for Locomotion. Journal of Applied Biomechanics 16(4): 419-427, 2000.
- [Background] van der Heeden JF, Marinus J, Martinez-Martin P, Rodriguez-Blazquez C, Geraedts VJ, van Hilten JJ. Postural instability and gait are associated with severity and prognosis of Parkinson disease. Neurology. 2016 Jun 14;86(24):2243-50. doi: 10.1212/WNL.0000000000002768. Epub 2016 May 13. PMID 27178702
- [Background] Cunnington R, Iansek R, Bradshaw JL, Phillips JG. Movement-related potentials in Parkinson's disease. Presence and predictability of temporal and spatial cues. Brain. 1995 Aug;118 ( Pt 4):935-50. doi: 10.1093/brain/118.4.935. PMID 7655889
- [Background] Morris ME, Iansek R, Matyas TA, Summers JJ. Stride length regulation in Parkinson's disease. Normalization strategies and underlying mechanisms. Brain. 1996 Apr;119 ( Pt 2):551-68. doi: 10.1093/brain/119.2.551. PMID 8800948
- [Background] Kestenbaum M, Fahn S. Safety of IPX066 , an extended release carbidopa-levodopa formulation, for the treatment of Parkinson's disease. Expert Opin Drug Saf. 2015 May;14(5):761-7. doi: 10.1517/14740338.2015.1015986. Epub 2015 Feb 19. PMID 25697185
- [Background] Oung QW, Muthusamy H, Lee HL, Basah SN, Yaacob S, Sarillee M, Lee CH. Technologies for Assessment of Motor Disorders in Parkinson's Disease: A Review. Sensors (Basel). 2015 Aug 31;15(9):21710-45. doi: 10.3390/s150921710. PMID 26404288
- [Background] Rochester L, Hetherington V, Jones D, Nieuwboer A, Willems AM, Kwakkel G, Van Wegen E. The effect of external rhythmic cues (auditory and visual) on walking during a functional task in homes of people with Parkinson's disease. Arch Phys Med Rehabil. 2005 May;86(5):999-1006. doi: 10.1016/j.apmr.2004.10.040. PMID 15895348
- [Background] del Olmo MF, Arias P, Furio MC, Pozo MA, Cudeiro J. Evaluation of the effect of training using auditory stimulation on rhythmic movement in Parkinsonian patients--a combined motor and [18F]-FDG PET study. Parkinsonism Relat Disord. 2006 Apr;12(3):155-64. doi: 10.1016/j.parkreldis.2005.11.002. Epub 2006 Feb 3. PMID 16459124
- [Background] Ford MP, Malone LA, Nyikos I, Yelisetty R, Bickel CS. Gait training with progressive external auditory cueing in persons with Parkinson's disease. Arch Phys Med Rehabil. 2010 Aug;91(8):1255-61. doi: 10.1016/j.apmr.2010.04.012. PMID 20684907
- [Background] Baker K, Rochester L, Nieuwboer A. The effect of cues on gait variability--reducing the attentional cost of walking in people with Parkinson's disease. Parkinsonism Relat Disord. 2008;14(4):314-20. doi: 10.1016/j.parkreldis.2007.09.008. Epub 2007 Nov 7. PMID 17988925
- [Background] Taborri J, Palermo E, Rossi S, Cappa P. Gait Partitioning Methods: A Systematic Review. Sensors (Basel). 2016 Jan 6;16(1):66. doi: 10.3390/s16010066. PMID 26751449
- [Background] Trojaniello D, Ravaschio A, Hausdorff JM, Cereatti A. Comparative assessment of different methods for the estimation of gait temporal parameters using a single inertial sensor: application to elderly, post-stroke, Parkinson's disease and Huntington's disease subjects. Gait Posture. 2015 Sep;42(3):310-6. doi: 10.1016/j.gaitpost.2015.06.008. Epub 2015 Jun 25. PMID 26163348
- [Background] Ozminkowski RJ, Wells TS, Hawkins K, Bhattarai GR, Martel CW, Yeh CS. Big Data, Little Data, and Care Coordination for Medicare Beneficiaries with Medigap Coverage. Big Data. 2015 Jun;3(2):114-25. doi: 10.1089/big.2014.0034. PMID 27447434
- [Background] Iosa M, Fusco A, Morone G, Pratesi L, Coiro P, Venturiero V, De Angelis D, Bragoni M, Paolucci S. Assessment of upper-body dynamic stability during walking in patients with subacute stroke. J Rehabil Res Dev. 2012;49(3):439-50. doi: 10.1682/jrrd.2011.03.0057. PMID 22773202
- [Background] Iosa M, Fusco A, Morone G, Paolucci S. Development and decline of upright gait stability. Front Aging Neurosci. 2014 Feb 5;6:14. doi: 10.3389/fnagi.2014.00014. eCollection 2014. PMID 24550829
- [Background] Iosa M, Morelli D, Marro T, Paolucci S, Fusco A. Ability and stability of running and walking in children with cerebral palsy. Neuropediatrics. 2013 Jun;44(3):147-54. doi: 10.1055/s-0033-1336016. Epub 2013 Mar 13. PMID 23487325
- [Background] Iosa M, Morone G, Fusco A, Marchetti F, Caltagirone C, Paolucci S, Peppe A. Loss of fractal gait harmony in Parkinson's Disease. Clin Neurophysiol. 2016 Feb;127(2):1540-1546. doi: 10.1016/j.clinph.2015.11.016. Epub 2015 Dec 2. PMID 26679417
- [Background] Iosa M, Morelli D, Nisi E, Sorbara C, Negrini S, Gentili P, Paolucci S, Fusco A. Assessment of upper body accelerations in young adults with intellectual disabilities while walking, running, and dual-task running. Hum Mov Sci. 2014 Apr;34:187-95. doi: 10.1016/j.humov.2014.02.005. Epub 2014 Mar 11. PMID 24630612
- [Background] Manns PJ, Baldwin E. Ambulatory activity of stroke survivors: measurement options for dose, intensity, and variability of activity. Stroke. 2009 Mar;40(3):864-7. doi: 10.1161/STROKEAHA.108.531590. Epub 2009 Jan 15. PMID 19150867
- [Background] Skidmore FM, Mackman CA, Pav B, Shulman LM, Garvan C, Macko RF, Heilman KM. Daily ambulatory activity levels in idiopathic Parkinson disease. J Rehabil Res Dev. 2008;45(9):1343-8. PMID 19319758
- [Background] Padua L, Pazzaglia C, Pareyson D, Schenone A, Aiello A, Fabrizi GM, Cavallaro T, Santoro L, Manganelli F, Gemignani F, Vitetta F, Quattrone A, Mazzeo A, Russo M, Vita G; CMT-TRIAAL Group. Novel outcome measures for Charcot-Marie-Tooth disease: validation and reliability of the 6-min walk test and StepWatch() Activity Monitor and identification of the walking features related to higher quality of life. Eur J Neurol. 2016 Aug;23(8):1343-50. doi: 10.1111/ene.13033. Epub 2016 May 10. PMID 27160471
- [Background] Mileti I, Germanotta M, Di Sipio E, Imbimbo I, Pacilli A, Erra C, Petracca M, Rossi S, Del Prete Z, Bentivoglio AR, Padua L, Palermo E. Measuring Gait Quality in Parkinson's Disease through Real-Time Gait Phase Recognition. Sensors (Basel). 2018 Mar 20;18(3):919. doi: 10.3390/s18030919. PMID 29558410